CLINICAL TRIAL: NCT03687398
Title: Comparison of Genomic Maps of Endometrial Tissues of Patients With Endometriosis and Healthy Controls Via Nanochannel Technique and Proteomic-genomic Analyzes.
Brief Title: Genomic Maps of Endometrial Tissues of Patients With Endometriosis and Healthy Controls
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Acibadem University (Other)
Responsible Party: Sponsor
Other Study IDs: AcibademU endo
Record Dates: First submitted 2018-09-16; First posted 2018-09-27 (Actual); Last update posted 2019-07-09 (Actual); Status verified 2019-07

CONDITIONS: Endometriosis; Endometrioma
Keywords: genetic analysis; endometriosis; nanoclonal; copy number
MeSH Terms: conditions — Endometriosis | interventions — Genetic Testing

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- control: does not have endometriosis or related diseases and not under any drug therapy does not have any benign or malign disease
  Interventions: Diagnostic Test: genetic testing with nanoclonal technique
- patient: has laparoscopically proven endometriosis
  Interventions: Diagnostic Test: genetic testing with nanoclonal technique

INTERVENTIONS:
Diagnostic Test: genetic testing with nanoclonal technique — endometrial sampling

SUMMARY:
Endometriosis is a chronic inflammatory disease that affects 10-17% of women in childbearing age, 35-60% of women with chronic pelvic pain and can cause infertility, costing as much as 2.8 billion dollars per year. For this reason, every step taken in diagnosis and treatment is of great importance both materially and spiritually. Patients can be diagnosed about 8-9 years after the onset of their complaints due to inadequacy of diagnostic methods In the study, it is decided to look at the basis of the disease, endometrial cells. And aimed to find the difference between the two women who are thought to be no different from each other among our current knowledge but one has endometriosis while other have not.

DETAILED DESCRIPTION:
Endometriosis is the appearance of a tissue similar to the endometrium in the ovaries, large intestine, and many other organ walls, except the uterus. The reason is unknown yet. Severe periodic pain, infertility, and pain during intercourse, affects approximately 2 million women in Turkey on average, 10% of women around the world. Endometriosis is a chronic inflammatory disease that affects 10-17% of women in childbearing age, 35-60% of women with chronic pelvic pain and can cause infertility, costing as much as 2.8 billion dollars per year. For this reason, every step taken in diagnosis and treatment is of great importance both materially and spiritually. Patients can be diagnosed about 8-9 years after the onset of their complaints due to the inadequacy of diagnostic methods In the study, it is decided to look at the basis of the disease, endometrial cells. And aimed to find the difference between the two women who are thought to be no different from each other among our current knowledge but one has endometriosis while others have not. For this reason, mapping of all genomes with the nanoclonal technique, the most advanced genetic screening method currently available from endometrial samples of patients and healthy women, is to identify the possible copy numbers, translocation, insertion and inversion anomalies, and to name them functionally by proteomic analysis. We believe that the results obtained from our study will guide the diagnostic tests and possible gene therapy in the future.

ELIGIBILITY:
Inclusion Criteria:

surgically diagnosed with endometriosis disease

* no diagnosıs for malignancy
* gave informed consent for application to the study enrolle as patient group females
* between 18-45 years old
* without any health conditions
* applied to the clinic for routine checkups for control group

Exclusion Criteria:

* being diagnosed with any kind of malignancy having trouble with endometrial cavity sampling

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — only seen in females
Study Population: patients who are :
  * surgically diagnosed with endometriosis disease
  * have no diagnosıs for malignancy
  * gave informed consent for application to the study enrolle as patient group
  females
  * between 18-45 years old
  * without any health conditions
  * applied to the clinic for routine checkups are going to be taken as the control group
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2018-10-01 (Actual); Primary Completion 2020-08-01 (Estimated); Study Completion 2020-09-01 (Estimated)

PRIMARY OUTCOMES:
diagnostic testing | 2 years
  finding a genetic difference which specifically preserved in endometriosis patients but not in healthy controls. To analyse the different region on chromosomes and name the pathophysiology underlying it

CONTACTS AND LOCATIONS:
Overall Officials: Bahar Yuksel, Study Director — md
Locations (1):
- Bahar Yuksel, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Cao H, Hastie AR, Cao D, Lam ET, Sun Y, Huang H, Liu X, Lin L, Andrews W, Chan S, Huang S, Tong X, Requa M, Anantharaman T, Krogh A, Yang H, Cao H, Xu X. Rapid detection of structural variation in a human genome using nanochannel-based genome mapping technology. Gigascience. 2014 Dec 30;3(1):34. doi: 10.1186/2047-217X-3-34. eCollection 2014. PMID 25671094
- [Result] Kobayashi H, Imanaka S, Nakamura H, Tsuji A. Understanding the role of epigenomic, genomic and genetic alterations in the development of endometriosis (review). Mol Med Rep. 2014 May;9(5):1483-505. doi: 10.3892/mmr.2014.2057. Epub 2014 Mar 14. PMID 24639062